CLINICAL TRIAL: NCT05609448
Title: Real-time MR Imaged Treatment With Holmium Microspheres of Patients With Primary Liver Cancer; a Single Center, Interventional, Non-randomized, Feasibility Study
Brief Title: MRI-guided Holmium-166 Radioembolization
Acronym: EMERITUS-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Radboud University Medical Center (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMERITUS-2
Record Dates: First submitted 2022-10-26; First posted 2022-11-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Primary Liver Cancer; Non-Resectable Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; radioembolization; TARE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-guided radioembolization (Experimental): Study patients will receive radioembolization with holmium microspheres in an MRI guided setting.
  Interventions: Procedure: MRI-guided radioembolization

INTERVENTIONS:
Procedure: MRI-guided radioembolization — Catheter placement will be performed using fluoroscopy, after which patients are transferred to the MRI scanner, where holmium microspheres are administered based on MRI dosimetry. Thereby, patients get a personalized dose administration.

SUMMARY:
To investigate the safety and feasibility of a personalized Ho-166-PLLA-MS TARE approach by using MRI guidance in inoperable patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hepatocellular carcinoma BCLC stage B or C
2. At least one lesion of 10 mm or more in the longest diameter on contrast-enhanced MRI/CT
3. Patient is eligible for TARE as determined by the tumour board (in Dutch: MDO)
4. Patient has a life expectancy of 12 weeks or longer
5. Patient has a WHO performance score of 0-2

Exclusion Criteria:

1. Extrahepatic disease that cannot be targeted during the TARE session (enlarged lymph nodes in the liver hilus are allowed)
2. Radiation therapy, chemotherapy or major surgery within 4 weeks before treatment
3. Serum bilirubin > 2.0 x the upper limit of normal
4. ALAT, ASAT, alkaline phosphatase (AF) > 5x the upper limit of normal
5. Leukocytes <4.0 * 109/L or platelet count <60 * 109/L
6. Significant heart disease that in the opinion of the physician increases the risk of ventricular arrhythmia.
7. Pregnancy or breast feeding
8. Disease with increased chance of liver toxicity, such as primary biliary cirrhosis or xeroderma pigmentosum
9. Patients ineligible to undergo MR-imaging (claustrophobia, metal implants, etc)
10. Portal vein thrombosis of the main branch (more distal branches are allowed)
11. Untreated, active hepatitis
12. Body weight > 150 kg (because of maximum table load)
13. Severe allergy for i.v. contrast (Iomeron, Dotarem and/or Primovist)
14. Lung shunt > 30 Gy, as calculated using scout dose 166Ho SPECT/CT.
15. Uncorrectable extrahepatic deposition of scout dose activity. Activity in the falciform ligament, portal lymph nodes or gallbladder are accepted.
16. Unstable final catheter position due to hepatic artery anatomy, which might lead to dislocation of the catheter during transfer to the MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of dose administration cohorts | 12 months after treatment
  Determine a safe maximal healthy liver dose for personalised administration of microspheres based on (S)AEs related to liver toxicity due to radioembolisation.
Safety of MRI-guided radioembolization procedure | 12 months after treatment
  Monitoring (S)AE's related to the investigated combination of MRI-guided 166Ho radioembolization.
Time constraints of performing intraprocedural MRI-based dosimetry | during treatment procedure
  Time constraints for image processing in between administration of microspheres, in order to be able to perform the procedure within half a day.
Feasibility of performing intraprocedural treatment planning | during treatment procedure
  The ability of deciding on catheter positions and dose aministration during the procedure based on MRI dosimetry by comparing the standard of care treatment plan to the treatment performed during the study.

SECONDARY OUTCOMES:
Dosimetry optimization | 12 months after treatment
  Perform optimization of holmium dosimetry using SPECT and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Frank Nijsen, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data is available to other researchers upon reasonable request